CLINICAL TRIAL: NCT01920997
Title: Qing'E Formula Therapy on Menopausal Symptoms (Healthy Volunteers Recruitment for Control Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QE-2458-3
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Healthy; normal menstrual cycles

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (1):
- No drug intervention: The objective of this study is to investigate the expression of NEI network and urine metabolomics of healthy women with normal menstrual cycles.

SUMMARY:
This study will recruit 50 healthy women with normal menstrual cycles aged 40-50, to investigate the expression of their NEI network and urine metabolomics.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women with normal menstrual cycles aged 40-50.
2. The score of Kupperman index is less than 15.
3. Not alcoholics or smokers (past or smoking).
4. Get subjects informed consent process should comply with GCP requirements.

Exclusion Criteria:

1. Volunteers with heart, liver, kidney disease or acute or chronic gastrointestinal diseases, or with diseases of blood, endocrine, neurological and other systems.
2. Volunteers are participating in other clinical trials within 3 months.
3. Volunteers who donated blood or loosed blood heavily within 3 months.
4. Volunteers with previous history of mental illness, drug abuse or drug dependence.
5. Volunteers who took drugs within 14 days before the trail.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women with normal menstrual cycles aged 40-50
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The expression of NEI network and Urine metabolomics | 2-5 days after menstruation
  The indices of NEI network include:
  1. Hypothalamic-pituitary-adrenal axis: CRH, ATCH, CORT
  2. Hypothalamic-pituitary-thyroid axis: TRH, T3, T4
  3. Renin - angiotensin - aldosterone system: PRA, Ang2, ALD
  4. Sex hormones: E2, FSH
  5. Immune factors: TNF-α、IL-6、IL-1
  6. Cardiovascular indicators: ET, NO, Hcy, Folic acid

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China